CLINICAL TRIAL: NCT02671279
Title: Effect of 6 Days Low Calorie Diet Before Bariatric Surgery
Brief Title: Low Calorie Diet in Morbidly Obese Patients
Acronym: PreBar
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Fonna (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2015/361
Record Dates: First submitted 2015-07-13; First posted 2016-02-02 (Estimated); Last update posted 2020-02-13 (Actual); Status verified 2017-12

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Low calorie diet (Other): Dietary intervention group
  Interventions: Dietary Supplement: Low calorie diet

INTERVENTIONS:
Dietary Supplement: Low calorie diet — 6 days of low calorie diet, estimated kcal 400-600/day.

SUMMARY:
This is a prospective study of morbidly obese patients that are planned to conduct bariatric surgery. The patients included in the study will conduct a low-calorie diet for 6 days prior to the operation and be admitted to hospital for this period. On admission and after finishing the diet a number of tests will be performed: Weigh, height, oral glucose tolerance test, bioimpedance measurement, and samples of blood, urine and a biopsy of subcutaneous adipose tissue.

DETAILED DESCRIPTION:
The study will include 14 patients planned for bariatric surgery with BMI 40-46. The patients will be admitted to hospital 8 days prior to planned surgery and conduct a diet based mostly on fluids (yogurt, soups). Estimated daily calorie intake will be 400-600 kcal.

At the day of admission and at day 7 a number of tests will be performed including blood tests, urine test and biometric measurement and a biopsy of subcutaneous adipose tissue. Weight will be measured every morning for the study period.

During the operation fatty tissue samples will be taken subcutaneous and from the omentum major.

This study is planned as a control group to another study where blood tests and subcutanous adipose tissue was sampled before and 6 days after bariatric surgery. The main aim of this study is to compare changes in adipose tissue and blood samples for patients before and 6 days after surgery to before and 6 days after a low-calorie diet.

ELIGIBILITY:
Inclusion Criteria:

* BMI 40-46 kg/m2
* The patients must not conduct a diet before admission.
* Fasting blood glucose <-7 nmol/l

Exclusion Criteria:

* Diabetes mellitus
* Treatment with antidiabetics
* Allergy for substances in the planned study-diet

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Changes in adipose gene expression signatures in obese subjects after 6 days of low-calorie diet | 8 days

SECONDARY OUTCOMES:
Changes in metabolomic signatures in obese subjects after 6 days of low-calorie diet | 8 days

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Mellgren, MD, PhD, Principal Investigator — Haukeland University Hospital
Locations (2):
- Norway (2):
  - Haukeland University Hospital, Bergen, Hordaland
  - Haugesund Sjukehus, Helse Fonna, Haugesund

IPD SHARING:
Plan to Share IPD: No